CLINICAL TRIAL: NCT05369962
Title: Adverse Event Prediction in Geriatric Patients in the ED With Ultrasound
Acronym: AGEDU
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Svenja Lichelle Haak, Principal Investigator, University Medical Center Groningen
Other Study IDs: 202100945
Record Dates: First submitted 2022-03-21; First posted 2022-05-11 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Adverse Event
MeSH Terms: conditions — Frailty | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Ultrasound measurements of the Qcsa

SUMMARY:
The aim of this study is to evaluate whether ultrasound measurements of the Qcsa can be utilized to identify older patients who are at risk for functional decline, ED revisit or death.

DETAILED DESCRIPTION:
Background:

Older people visit the Emergency Department (ED) more frequently then younger people and have a higher risk of functional decline, ED revisit or death. Several screening tools (such as the Dutch safety management system (VMS) and Acutely Presenting Older Patient (APOP)) have been developed to identify patients at the highest risk of adverse outcomes. Almost all require adequate communication with the patient, which is not always possible, for example when elderly patients present with a delirium. Point of Care Ultrasonography (POCUS) may be a valuable alternative screening tool in these instances.

Main research question:

To identify whether POCUS measurement of the rectus femoris muscle cross-sectional area (Qcsa) can be used as an alternative screening tool to predict functional decline, ED revisit or death in elderly patients in the ED.

Design (including population, confounders/outcomes):

This is a single centre prospective trial. Patients >70 years and older presenting in the ED of the University Medical Centre Groningen (UMCG) who are participating in the Acutelines bio-databank are eligible for inclusion. 68 patients will be included. Data will be extracted from the Acutelines bio-databank. A trained physician will perform ultrasound measurements in a standardized way.

Expected results:

The aim of this study is to evaluate whether ultrasound measurements of the Qcsa can be utilized to identify older patients who are at risk for functional decline, ED revisit or death.

ELIGIBILITY:
Inclusion Criteria:

* Age (>70 years)
* Presenting to the ED of the UMCG for one of the following specialties: internal medicine, nephrology, geriatric medicine, oncology, hematology, lung medicine, gastrointestinal/liver medicine, or emergency medicine (non-trauma).
* Consent obtained for participation in the Acutelines bio-databank

Exclusion Criteria:

* Unable to obtain ultrasound image of rectus femoris (e.g. amputation, edema)
* Paresis or paralysis of one or both legs

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients >70 years and older presenting in the ED of the UMCG hospital who are participating in the Acutelines bio-databank are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Ultrasound Qcsa | 1 day of admission to ED
  POCUS Qcsa in older patients in the ED.
ED revisit | 3 months
  Is there a relation between the performed POCUS Qcsa measurement at ED visit and ED revisit in older patients.
Mortality | 3 months
  Is there a relation between the performed POCUS Qcsa measurement at ED visit and mortality in older patients.

SECONDARY OUTCOMES:
ED revisit: Ultrasound Qcsa versus Karnofsky Performance Score | 3 months
  To compare the ability of the Qcsa ultrasound versus the Karnofsky Performance Score (gold standard) to predict ED revisit in older patients in the ED.
Mortality: Ultrasound Qcsa versus Karnofsky Performance Score | 3 months
  To compare the ability of the Qcsa ultrasound versus the Karnofsky Performance Score (gold standard) to predict mortality in older patients in the ED.
ED revisit: Ultrasound Qcsa plus Karnofsky Performance Score | 3 months
  To compare the added value of Qcsa ultrasound versus the Karnofsky Performance Score (gold standard) to predict ED revisit in older patients in the ED.
Mortality: Ultrasound Qcsa plus Karnofsky Performance Score | 3 months
  To compare the added value of Qcsa ultrasound versus the Karnofsky Performance Score (gold standard) to predict mortality in older patients in the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Haak, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT05369962/Prot_SAP_000.pdf